CLINICAL TRIAL: NCT05639933
Title: A Randomized, Placebo-controlled, Parallel Phase 2a Dose-ranging Study to Investigate the Efficacy, Safety, and Tolerability of Topical HT-001 for the Treatment of Skin Toxicities Associated With Epidermal Growth Factor Receptor Inhibitors
Brief Title: Study to Investigate the Efficacy, Safety, and Tolerability of Topical HT-001 for the Treatment of Skin Toxicities Associated With Epidermal Growth Factor Receptor Inhibitors
Acronym: CLEER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoth Therapeutics, Inc. (Other)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CLEER-001
Record Dates: First submitted 2022-11-14; First posted 2022-12-07 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Acneiform Eruption Due to Chemical; Xerosis Cutis; Paronychia
Keywords: Acneiform rash; EGFR inhibitor; Cutaneous toxicities
MeSH Terms: conditions — Paronychia | interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Open-Label PK Cohort (Experimental): Topical treatment with HT-001 2% Gel unblinded.
  Interventions: Drug: HT-001 2% Topical Gel
- Randomized, Double Blind Cohort (Placebo Comparator): Topical treatment with HT-001 (2%, 1%, or 0.5%) or placebo (HT-001 vehicle), blinded
  Interventions: Drug: HT-001 2% Topical Gel; Drug: HT-001 1% Topical Gel; Drug: HT-001 0.5% Topical Gel; Drug: HT-001 Placebo

INTERVENTIONS:
Drug: HT-001 2% Topical Gel — Topical gel, 2% active
Drug: HT-001 1% Topical Gel — Topical gel, 1% active
  Arms: Randomized, Double Blind Cohort
Drug: HT-001 0.5% Topical Gel — Topical gel, 0.5% active
  Arms: Randomized, Double Blind Cohort
Drug: HT-001 Placebo — Topical gel, vehicle gel
  Arms: Randomized, Double Blind Cohort

SUMMARY:
The goal of this clinical trial is to learn about HT-001 Topical Gel for treatment of EGFR inhibitor-induced skin toxicities. The main questions it aims to answer are:

* Determine the therapeutic effect of HT-001 for treatment of patients who develop acneiform rash undergoing Epidermal Growth Factor inhibitor (EGFRI) therapy using the acneiform rash investigator's global assessment scale [ARIGA]
* Evaluate the safety of HT-001 during treatment

Participants will apply HT-001 Gel once per day for 6 weeks, during which the effect on treating acneiform rash or other skin disorders induced by EGFRI therapy will be evaluated using different assessment tools to measure severity of rash, pain, and itching (pruritus), as well as the change in quality of life.

The study will be completed in 2 periods: the first period is open-label (unblinded) and all patients will receive HT-001 topical gel with the active ingredient; the second period is blinded and patients will be randomized to receive one of three concentrations of HT-001 or placebo.

Researchers will compare HT-001 to the placebo in the second period to see if HT-001 provides a significant treatment effect.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multi-center Phase 2a dose-ranging study to evaluate the efficacy, safety, and tolerability of HT-001 for treatment of EGFRI-induced skin toxicity. The study will include adult patients (≥ 18 years of age) scheduled to receive initial or repeat EGFRI therapy.

The study will be conducted in 2 periods: Part 1, an open-label cohort consisting of 12 patients to measure pharmacokinetics of HT 001 gel followed by Part 2, a randomized, parallel arm study comparing 3 dose strengths of HT-001 gel to placebo (HT 001 vehicle). Patients in the randomized cohorts will be randomly assigned to 1 of the 4 treatment arms in a 2:2:2:1 ratio (active groups = 2: placebo = 1).

All patients in both open-label and blinded cohorts will apply the study drug once a day to each area affected with cutaneous toxicity up to 30% body surface area (BSA) involvement, inclusive of skin, scalp, and nails.

The goal of the study is to determine the minimum efficacious dose strength(s) for further investigation. The dose effect, together with the application site safety assessments, and therapeutic effects based on the primary and secondary endpoints will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient (ie, ≥ 18 years of age at Screening/Baseline [V1]) prescribed an approved EGFRI to treat cancer (indication within the approved labeling for the EGFRI).
2. Patient has developed a rash or symptoms of a rash (papular and/or pustular eruptions) or symptoms of a rash (cutaneous burning), as assessed by both Common Terminology Criteria for Adverse Events (CTCAE) grading and ARIGA scales (severity

   ≤ 3) with overall involvement ≤ 30% BSA.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
4. Predicted life expectancy ≥ 3 months.
5. Patient is able and willing to comply with contraceptive requirements.
6. Patient must have the ability and willingness to attend the necessary visits (telehealth and in person).
7. Patient must be willing and able to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures.

Exclusion Criteria:

1. Patient has severe cutaneous toxicity (severity = 4 on the CTCAE grading and ARIGA scales) or cutaneous toxicity involvement that is > 30% BSA, or other severe systemic toxicity (severity > 3 on the CTCAE v5.0 scale) as a result of EGFRI therapy.
2. Patient has any underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the patient would comply with the protocol or complete the study per protocol.
3. Patient has a history of other skin disorders (eg, atopic dermatitis, psoriasis, recurrent skin infections), or history of illness that, in the opinion of the Investigator, would confound results of the study or pose unwarranted risk in administering study drug to the patient.
4. Patient has abnormal laboratory values at Screening/Baseline (V1):

   1. Absolute neutrophil count < 1000/mm3 and WBC count < 3000/mm3
   2. Platelet count < 50,000/mm3
   3. Aspartate transaminase (AST) > 2.5 × upper limit of normal (ULN)
   4. Alanine transaminase (ALT) > 2.5 × ULN
   5. Bilirubin > 1.5 × ULN
   6. Creatinine > 1.5 × ULN
5. Patient has a prescribed cancer treatment plan that requires radiation treatment to the head, neck, or upper trunk concurrent with EGFRI therapy or has previously received radiation therapy within 4 weeks prior to Screening/Baseline (V1).
6. Patient has received aprepitant or other neurokinin-1 receptor antagonist within 4 weeks prior to Screening/Baseline (V1).
7. Patient has had prior treatment with an investigational drug within 4 weeks prior to Screening/Baseline (V1), or at least 8 half-lives of the drug, whichever is longer.
8. Patient has an active infection (eg, pneumonia) or any uncontrolled disease except for the malignancy that, in the opinion of the Investigator, might confound the result or the study or pose unwarranted risk in administering the study drug to the patient.
9. Patient has received non-stable escalating doses of topical antibiotics, topical steroids, or other topical treatments within 14 days prior to Screening/Baseline (V1). Patients who have been on stable doses of topical antibiotics, topical steroids, or other topical treatments for 14 days or more are allowed to be enrolled and to stay on their current prescription. Reduction in dose due to improvement in EGFRI-related toxicities is allowed.
10. Patient has used non-stable escalating doses of systemic steroids within 14 days prior to Screening/Baseline (V1) excluding low-dose systemic corticosteroids as part of standard of care for prevention or treatment of chemotherapy-induced nausea and vomiting; acceptability of the steroid and dose is to be determined by the study Investigator. Patients who have been on a stable dose of systemic steroids for 14 days or more are allowed to be enrolled and to stay on their current prescription. Reduction in dose due to improvement in EGFRI-related toxicities is allowed. Use of steroid inhalers and nasal corticosteroids is allowed.
11. Patient has received non-stable escalating dose treatment with a systemic antibiotic within 14 days prior to Screening/Baseline (V1). Patients who have been on stable doses of systemic antibiotics for 14 days or more are allowed to be enrolled and to stay on their current prescription. Reduction in dose due to improvement in EGFRI-related toxicities is allowed.
12. Patient has received concomitant treatment with pimozide, moderate to strong cytochrome p450 (CYP) 3A4 inhibitors (diltiazem, ketoconazole, itraconazole, nefazodone, troleandomycin, clarithromycin, ritonavir, nelfinavir), or strong CYP3A4 inducers (rifampin, carbamazepine, phenytoin) within 30 days of Screening/Baseline (V1).
13. Patient has a history of hypersensitivity to aprepitant or any component of HT-001.
14. Patient is pregnant or lactating at Screening/Baseline (V1) or planning to become pregnant (self or partner) at any time during the study, including the follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Acneiform Rash Investigator's Global Assessment Scale [ARIGA ] | 6 weeks
  Proportion of patients with a grade ≤ 1 based on the Acneiform Rash Investigator's Global Assessment [ARIGA] Scale; novel 5-point scale 0-4 with score of 0 is clear and grade 4 being most severe
Pharmacokinetics of HT-001 applied topically [Cohort 1] - Area Under the Curve (AUC) | Day 1 and Day 42
  Characterize pharmacokinetics of HT-001 parameters including: measured drug concentrations above the lower limit of quantitation, number of patients with measurable systemic exposure; if data allow - area under the curve (AUC)
Pharmacokinetics of HT-001 applied topically [Cohort 1] - Peak Plasma Concentration (Cmax) | Day 1 and Day 42
  Characterize pharmacokinetics of HT-001 parameters including: maximum (or peak) serum concentration (Cmax)

SECONDARY OUTCOMES:
Pruritus Numeric Rating Scale (NRS) | 3 weeks and 6 weeks
  Change from Baseline in Pruritus Numeric Rating Scale (average itch and worst itch); The numerical scale is ranked from 0 ("no itch") to 10 ("worst imaginable itch").
Pain Numeric Rating Scale | 3 weeks and 6 weeks
  Change from Baseline in pain based on a 11-point NRS (where "0" indicates "no pain", "5" indicates "moderate pain" and "10" indicates "worst pain imaginable")
Change in acneiform rash severity | 3 weeks and 6 weeks
  Change from Baseline in acneiform rash grade based on the Acneiform Rash Investigator's Global Assessment Scale [ARIGA]; novel 5-point scale 0-4 with score of 0 is clear and grade 4 being most severe
Time to improvement | 6 weeks Day 1- Day 42
  Time to improvement in at least one grade using the Acneiform Rash Investigator's Global Assessment Scale [ARIGA ] for acneiform rash; novel 5-point scale 0-4 with score of 0 is clear and grade 4 being most severe
Time to rescue therapy | Treatment Day 1- Day 42
  Time to topical rescue therapy treatment after initiation of HT-001
EGFR Inhibitor dose reduction or discontinuation | Treatment Day 1- Day 42
  Proportion of patients with EGFRI dose reduction or discontinuation during the 6-week treatment period
Safety and tolerability of HT-001 | screening, Day 1 - 42, follow-up (Day 56)
  Incidence of treatment-emergent adverse events and treatment-emergent serious adverse events
Modified Draize Scale | Day 1, 7, 21, 35, 42, 56
  Assessment of skin irritation through measurement of cutaneous signs of erythema (score 0-3; 3 is most severe) and edema (add 0.5 if present)
Physical Examination | Day 1, 7, 21, 35, 42, 56
  full physical examination will include examination of general appearance, skin, neck (including thyroid), eyes, ears, nose, throat, heart, lungs, abdomen, lymph nodes, extremities, and nervous system. An AE form must be completed for all changes identified as clinically noteworthy.
Height | Screening
  Height recorded in inches
Body weight | Day 1, 21, 42, 56
  Body weight in pounds.

OTHER OUTCOMES:
Scoring system for paronychia related to oncologic treatments (SPOT) | Day 1, 7, 21, 35, 42
  Proportion of patients with improvement in paronychia based on the SPOT scale. Each parameter of paronychia, such as redness (R), edema (E), discharge (D) and granulation tissue (G), is evaluated on a 4-point scale from 0 to 3. The highest score for each R-E-D-G parameter among all involved fingers (or toes) of the respective hand (or foot) represents the overall score for that parameter on that hand (or foot) - note, the highest scores for the different parameters could originate from different fingers (or toes).
Xerosis Severity Scale | Day 1, 7, 21, 35, 42
  Proportion of patients with improvement in xerosis using the Xerosis Severity Scale adapted from Guenther et al. (Guenther et al., 2012). The assessment uses signs and symptoms of xerosis (such as rough/scaling skin, itching, pain, erythema, and fissures) as a composite score to determine the severity classification. In this scale, "-" indicates not present; "+"indicates a mild symptom; "++" indicates a moderate symptom; and "+++" indicates a severe symptom
Change in Quality of Life (QoL) | Day 1, 21, 42
  Change in quality of life based on FACT-EGFR-18. This 18-item QoL assessment was developed by Wagner et al. using a 5-point Likert scale (ie, 0 = not at all, 1 = a little bit, 2 = somewhat, 3 = quite a bit, and 4 = very much) with a recall period of the past 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Mario Lacouture, MD, Study Chair — NYU Langone Health
Locations (8):
- United States (8):
  - UCI Health - CIACC, Irvine, California
  - UC Irvine - Chao Family Cancer Center, Orange, California
  - The George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - NYU Langone Health, Mineola, New York
  - Northwell Physician Partners Dermatology, New Hyde Park, New York
  - Montefiore Medical Center, The Bronx, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guenther L, Lynde CW, Andriessen A, Barankin B, Goldstein E, Skotnicki SP, Gupta SN, Choi KL, Rosen N, Shapiro L, Sloan K. Pathway to dry skin prevention and treatment. J Cutan Med Surg. 2012 Jan-Feb;16(1):23-31. doi: 10.1177/120347541201600106. PMID 22417992